CLINICAL TRIAL: NCT05204485
Title: Prospective, Randomized-Control Trial Comparing Intramedullary Fibular Fixation With Standard Open Reduction And Internal Fixation In Diabetic Patients With Unstable Ankle Fracture
Brief Title: Diabetic Fibular Nail Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment making completion of the study impossible, relocation of both the PI and Co-PI
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB21-1218
Record Dates: First submitted 2022-01-12; First posted 2022-01-24 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Ankle Fractures
MeSH Terms: conditions — Ankle Fractures | interventions — Open Fracture Reduction; Fracture Fixation, Internal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fibular intramedullary nail (Active Comparator): Randomized in the OR to ankle fracture repair with fibular intramedullary nail
  Interventions: Procedure: Fibular intramedullary nail
- Open reduction and internal fixation (ORIF) (Active Comparator): Randomized in the OR to ankle fracture repair with ORIF
  Interventions: Procedure: Open reduction and internal fixation

INTERVENTIONS:
Procedure: Fibular intramedullary nail — The standard manufacturers approved technique will be performed including the use of 2 distal interlocking screws and the use of a minimum of 1 fibula pro tibia fixation screw depending on the patients' anatomical characteristics.
  Arms: Fibular intramedullary nail
Procedure: Open reduction and internal fixation — An open approach (direct lateral or posterolateral incision) will be carried out. The reduction will be performed using standard techniques of clamping and traction. Fixation will be performed after reduction of the fracture with a plate and screw construct. The surgeon will then proceed to perform surgical fixation of other associated fractures or ligament injuries as indicated. This will most often include open reduction and internal fixation of the medial malleolus with screws through a separate medial incision.
  Arms: Open reduction and internal fixation (ORIF)

SUMMARY:
Our null hypothesis is that fibular intramedullary fixation (IMFN) does not impact complication rates when compared to standard of care treatment with open reduction and internal fixation (ORIF). There are no current or past RCTs comparing these fixation techniques to one another in diabetic patients. There is good data supporting both the use of intramedullary fixation for fibular fractures alone, and in high-risk patient populations (elderly, and diabetics). However, the effectiveness of these methods with respect to each other has never been investigated. The knowledge gained will allow us to potentially influence and adapt protocols to treat this patient population. Additionally, resources available at our institution provide a supportive framework with which to maintain contact with patients after hospital discharge. These key factors will allow us to perform a robust analysis of this population, to include outcomes measures of function and complications.

DETAILED DESCRIPTION:
Our null hypothesis is that fibular intramedullary fixation (IMFN) does not impact complication rates when compared to standard of care treatment with open reduction and internal fixation (ORIF). There are no current or past RCTs comparing these fixation techniques to one another in diabetic patients. There is good data supporting both the use of intramedullary fixation for fibular fractures alone, and in high-risk patient populations (elderly, and diabetics). However, the effectiveness of these methods with respect to each other has never been investigated. The knowledge gained will allow us to potentially influence and adapt protocols to treat this patient population. Additionally, resources available at our institution provide a supportive framework with which to maintain contact with patients after hospital discharge. These key factors will allow us to perform a robust analysis of this population, to include outcomes measures of function and complications.

With much of the existing literature on fibular nails being retrospective with limited focus on the diabetic population, there is no clear guidance on when the use of this device is indicated. Retrospective studies in fracture patients bring in significant bias given that a specific surgical technique may be chosen because of individual patient factors including soft tissue condition, fracture pattern and perceived level of risk. This limits our understanding of how an implant will perform across the population of interest. Our approach to randomize our patients will reduce the bias that exists in the current literature. In addition, the only prospective study that has been performed on the fibular nail was in elderly patients in which only two patients were diabetic. Given the many challenges with high rates of infection in this patient population we seek intramedullary fibular fracture fixation as a treatment that could potentially change this existing paradigm

Primary Objective Compare post-operative all cause complications in diabetic patients with ankle fractures.

Secondary Objective(s) Compare patient reported outcomes, range of motion, pain and radiographic outcomes in patients treated with ORIF vs. fibular intramedullary nails.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Unstable ankle fracture
* Diagnosis of Diabetes:

  * Fasting BG > 120
  * Non-fasting BG > 200
  * HbA1c > 6.5

Exclusion Criteria:

* Patients not meeting inclusion criteria (stable fracture patterns, non-diabetics)
* Poly-trauma patients (multiple [>2] extremity injuries that interfere and/or limit patient mobilization
* Open fractures
* Delayed presentation of fracture (>4 weeks)
* Fractures that the treating surgeon indicates requires a posterior approach to achieve stability
* Patients with an active infection or wound at the ankle
* Utilizing worker's compensation at the time of screening
* Any previous ligament or fracture surgery on the index ankle
* Inflammatory rheumatic disease or other rheumatic disease
* Immune compromised patients (hepatitis, HIV, etc.)
* Non-English speaking patients
* Unwilling or unable to follow study protocol

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2024-01-19 (Actual); Study Completion 2024-01-19 (Actual)

PRIMARY OUTCOMES:
Composite complication rate | 1 year post-operatively
  The difference in overall composite complication rate between Fibular intramedullary fixation and ORIF

SECONDARY OUTCOMES:
Patient reported outcome scores | 1 year post-operatively
  Any difference in Patient reported outcomes scores (PROMIS Physical Function or Pain Interference CAT) score between Fibular Intramedullary fixation and ORIF

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Hynes, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers.